CLINICAL TRIAL: NCT03700268
Title: Programming Cochlear Implant With Artificial Intelligence
Acronym: CI_AI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017/04SEP/427; 2017/13OCT/480 (Other: CEHF of Cliniques Universitaires Saint Luc)
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Deafness; Perception
Keywords: Deafness; cochlear implant; Artificial Intelligence
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual fitting (Experimental): The patient is receiving the classical treatment : 10 sessions of 1 hour during one year where the clinician programs manually the Cochlear implant.
  Interventions: Other: Manual intervention to programme Cochlear Implant electrodes
- Artificial Intelligence (Experimental): The patient is receiving the new treatment : 4 sessions of 1 hour during one year where the clinician programs the Cochlear implant with the FOX (Fitting to Outcome eXpert) software using artificial intelligence.
  Interventions: Other: Manual intervention to programme Cochlear Implant electrodes

INTERVENTIONS:
Other: Manual intervention to programme Cochlear Implant electrodes — The Clinician test the 22 electrodes so that the patient is able to hear the language

SUMMARY:
This thesis project proposes to investigate the "state of the art" of the programming of the cochlear implant. In the center of audiophonologie Brussels, the classic 'manual programming' has been in use over 20 years and also the new way 'Artificial Intelligence programming'. The investigators want to compare, objectify, and control this new mode of programming.

The study is planned over 4 years, in order to test, randomized, 15 subjects with manual programming and 15 other subjects with Artificial Intelligence programming. To test the performance of Cochlear Implant patients, audiological, language auditory perception and questionnaire tests will be presented.

This research aims to determine the contribution and results of Artificial Intelligence programming.

ELIGIBILITY:
Inclusion Criteria:

* unilateral cochlear implant
* post-lingual hearing loss
* a good command of French.

Exclusion Criteria:

* non deaf
* bilateral cochlear implant
* deaf without cochlear implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Evaluate Fox software efficiency | 1 year
  Evaluate Fox software efficiency for the programming of Cochlear implants used to facilitate hearing of deaf patients. This research aims to determine the contribution (time, results,…) of Artificial intelligence to program cochlear implants. The investigator will compare the results of hearing tests of newly programmed patients with FOX to those of newly programmed patients with a manual fitting.
  The outcomes used by software FOX are pure tone audiometry thresholds from 250 to 6000Hz, speech audiometry scores at 40, 55, 70 and 85 dB SPL, spectral discrimination scores using an oddity test in which 2 speech sounds are presented and where the aim is to react to the odd speech sound (Govaerts et al. 2006), and loudness growth curves determined with narrow band noises centered at 250, 1000 and 4000 Hz using an A§E® test battery (Meeuws et al., 2017).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wathour J, Govaerts PJ, Lacroix E, Naima D. Effect of a CI Programming Fitting Tool with Artificial Intelligence in Experienced Cochlear Implant Patients. Otol Neurotol. 2023 Mar 1;44(3):209-215. doi: 10.1097/MAO.0000000000003810. Epub 2023 Jan 18. PMID 36728126
- [Derived] Wathour J, Govaerts PJ, Deggouj N. Variability of fitting parameters across cochlear implant centres. Eur Arch Otorhinolaryngol. 2021 Dec;278(12):4671-4679. doi: 10.1007/s00405-020-06572-w. Epub 2021 Jan 3. PMID 33388985
- [Derived] Wathour J, Govaerts PJ, Deggouj N. From manual to artificial intelligence fitting: Two cochlear implant case studies. Cochlear Implants Int. 2020 Sep;21(5):299-305. doi: 10.1080/14670100.2019.1667574. Epub 2019 Sep 17. PMID 31530099